CLINICAL TRIAL: NCT06538220
Title: Evaluation of the Care Pathway Offered by the "Chonic Disease Unit" to Obese Patients
Brief Title: Evaluation of the Care Pathway Offered by the "Chronic Disease Unit" to Obese Patients
Acronym: EVAMMACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Maison de la Maladie Chronique (Unknown); Institut d'Etude de la Maladie Chronique (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-CHITS-004; 2024-A00145-42 (Other: ID-RCB number)
Record Dates: First submitted 2024-07-26; First posted 2024-08-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Obesity
Keywords: Care pathway; Self-efficacy; Patient education; Obesity; Interdisciplinary; Self mangement
MeSH Terms: conditions — Obesity | interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obese patients (Experimental): Patients suffering from obesity defined by a BMI ≥ 30 and following the Chronic Disease Unit care pathway
  Interventions: Behavioral: Questionnaires and focus group

INTERVENTIONS:
Behavioral: Questionnaires and focus group — To evaluate the Chronic Disease Unit care pathway, patients will respond to questionnaires : quality of life (SF-12), personal efficacy scale (GSES), "Specific self Efficacy related to Weight Management" (SEWM), Rosenberg self-esteem, body image satisfaction (QIC), state of anxiety and depression (HAD), Chronic Disease Unit satisfaction. Some patients will also participate to focus group.

SUMMARY:
Obesity is a chronic and progressive disease medically defined as an increase in body fat, with consequences for physical, psychological and social well-being. With an estimated prevalence of 17% in France, obesity and its management remain a major public health issue. Projections by the World Health Organisation (WHO) show that the prevalence of non-communicable diseases, including obesity, is set to rise again by 2030 in all European countries.

To support patients and prevent obesity development, the French National Authority for Health (HAS) advocates change in practices and places patient education at the heart of care. The management of chronic diseases such as obesity must be offered on a long-term basis, adapting to complications onset, and patients must become active players in their treatment and the proposed care pathway. However, our experience shows that patients have difficulty finding their way around a care pathway and identifying the medical or paramedical resources that could help them to set their health goals and initiate change.

That's why the Var region has developed the "Chronic Disease Unit", which offers coordinated, adapted and individualised care pathways for patients suffering from chronic illnesses, including obesity; therapeutic education and the psychosocial dimension are at the heart of the Chronic Disease Unit approach. Depending on their psychosocial skills, each patient will be encouraged to develop skills at their own pace, but also to become autonomous in managing their illness and taking part in the healthcare decisions about them. To be autonomous, a patient must not only know what to do, but also feel able to do it, i.e. develop a sense of self-efficacy. When they have the necessary skills and believe in their abilities, patients are more likely to adopt health-promoting behaviours. While obesity generally seems to be linked to a low self-efficacy, the self-efficacy appears to be involved in weight management quality, commitment to a programme and the weight loss extent that results.

The aim of EVAMMACH study is to evaluate if the Chronic Disease Unit care pathway could promote obese patients' sense of self-efficacy and meet their expectations.

DETAILED DESCRIPTION:
Patients will be identified at the Chronic Disease Unit during an orientation consultation with the dietician as part of routine practice. The clinician, who is also the study investigator, will then select patients who meet the protocol's inclusion criteria and inform them of the research. He will explain the study in detail and give them the information letter.

Patients will then be seen again in consultation during 3 visits:

* M0: During this consultation, the investigating physician will obtain oral consent of patients to their participation in the research, resulting in a research consultation lasting around 45 minutes and including questionnaires completion: quality of life (SF-12), personal efficacy scale (GSES), "Specific self Efficacy related to Weight Management" (SEWM), Rosenberg self-esteem, body image satisfaction (QIC), state of anxiety and depression (HAD).
* M3: Follow-up visit with completion of SF-12, GSES, Rosenberg and QIC questionnaires.
* M6: Follow-up visit with completion of the same questionnaires as at M0 plus the Chronic Disease Unit satisfaction questionnaire, and end of research.

Questionnaires will be completed in presence of the Chronic Disease Unit psychologist, to offer a discussion or treatment if necessary.

During M0 and M6 visits, some patients will participate in a focus group. An audio recording of the focus group sessions will be made after obtaining the participants' consent.

ELIGIBILITY:
Inclusion Criteria:

1. Patient identified by the network or referred by a healthcare professional,
2. Patient aged 18 or over,
3. Patient suffering from obesity defined by a BMI ≥ 30,
4. Patient who understands and speaks French.

Exclusion Criteria:

1. Opposition of the patient to participation in the study,
2. Pregnant, parturient or breast-feeding woman,
3. Patient undergoing bariatric surgery,
4. Patient under judicial protection (guardianship, curatorship, etc.) or safeguard of justice,
5. Patients with unstable psychiatric disorders,
6. Patients on neuroleptics,
7. Any other reason which in the opinion of the investigator, could interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether the care pathway proposed by the Chronic Disease Unit improves the self-efficacy of obese patients at M6 | 0 month and 6 months (M6)
  The self-efficacy will be determined by the overall score obtained on the General Self-Efficacy Scale (GSES)
  [10;40] A high score corresponds to important self efficacy

SECONDARY OUTCOMES:
To evaluate whether the care pathway proposed by the Chronic Disease Unit improves the self-efficacy of obese patients at M3 | 0 month and 6 months (M6)
  The self-efficacy will be determined by the overall score obtained on the General Self-Efficacy Scale (GSES)
  [10;40] A high score corresponds to important self efficacy
To assess whether the care pathway improves overall quality of life at M3 and M6 | 0 month, 3 and 6 months
  The quality of life will be determined by the overall score obtained on the quality of life SF-12 questionnaire
  [0;100] A high score corresponds to better health/quality of life
Evaluate the effect of the treatment pathway on the patient's corpulence between M0 and M6. | 0 month and 6 months
  The patient's corpulence will be determined by BMI
To assess disruptions in care | 6 months
  Number of premature study exits and their causes
To study the socio-demographic and clinical characteristics of patients at M0 | 0 month
  Descriptive statistical analyses of socio-demographic and clinical characteristics at M0:
  * Socio-demographic data: age, sex, family and professional situation, education level, social disadvantage index.
  * Clinical data relating to obesity: existence of a known eating disorders or SCOFF score (eating disorders screening questionnaire), co-morbidities (diabetes, heart failure, obsessive-compulsive symptoms), BMI, diets followed, maximum and minimum weight achieved, etc.
  * Patient history: trauma, notorious violence and family history
  * Type of address (profession, town/city/network)
  * Current treatments: antidepressant, anxiolytic, etc.
  * Regular physical activity
  * Completion of ETP Obsession programme
Evaluate the effect of the Chronic Disease Unit care pathway between M0 and M6, in the subgroup of patients with Eating Disorders. | 0 month and 6 months
  Number of compulsive binges per week assessed in the subgroup of patients with eating disorders.
Evaluate patient adherence to the Chronic Disease Unit care pathway at M3 and M6 | 3 and 6 months
  The number of workshops/consultations carried out over the number of workshops/consultations planned in the patient's objectives using the ETP Pilote software at M3 and M6.
Assess patients' self-esteem at M0, M3 and M6 | 0 month, 3 and 6 months
  The patients' self-esteem will be determined by the score obtained on Rosenberg self-esteem scale
  [10;40] A high score corresponds to high self-esteem
Evaluate patient satisfaction with body image at M0, M3 and M6 | 0 month, 3 and 6 months
  The patient satisfaction with body image will be determined by the score of body image satisfaction (QIC) questionnaire
  [19;95] A high score corresponds to very good body satisfaction
Assess patients' anxiety and depression at M0 and M6 | 0 month and 6 months
  The patients' anxiety and depression level will be determined by the score of state of anxiety and depression (HAD) scale
  [0;42] A high score corresponds to anxiety or depressive disorders presents
Evaluate patient satisfaction with the Chronic Disease Unit care pathway at M6 | 6 months
  Patient satisfaction will be determined by the responses of the Chronic Disease Unit satisfaction questionnaire [0 : not at all satisfied;10 : completely satisfied]

OTHER OUTCOMES:
To assess whether the care pathway proposed by Chronic Disease Unit improves obese patients' sense of self-efficacy between M0 and M6. | 0 month and 6 months
  The self-efficacy will be determined by the overall score obtained on "Specific self Efficacy related to Weight Management (SEWM) questionnaire
  [0;400] A high score corresponds to a high sense of self-efficacy
Using the focus group method, to qualitatively assess the obese patient's experience before (M0) and after (M6) treatment in the Chronic Disease Unit care pathway. | 0 month and 6 months
  Qualitative analysis of recorded focus group

CONTACTS AND LOCATIONS:
Overall Officials: Aurelie GAZAGNE, Dietician, Study Director — MMC / IEMC
Locations (1):
- MMC, La Garde, Var, France

IPD SHARING:
Plan to Share IPD: No